CLINICAL TRIAL: NCT07322263
Title: Intravesical Gemcitabine and Docetaxel for High-Risk, BCG-Unresponsive Non-Muscle Invasive Bladder Cancer: A Prospective Cohort Study (GEMDOCE-BU)
Brief Title: Intravesical GEM/DOCE for HR BCG-Unresponsive NMIBC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Michael A. O'Donnell (Other)
Responsible Party: Sponsor-Investigator, Michael A. O'Donnell, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202508227
Record Dates: First submitted 2025-12-01; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-10

CONDITIONS: Bladder Cancer; Non-Muscle Invasive Bladder Cancer (NMIBC); Urothelial Carcinoma; Carcinoma in Situ (CIS); High-Grade Papillary Bladder Tumors; BCG-Unresponsive Bladder Cancer; Ta Stage Bladder Cancer; T1 Stage Bladder Cancer; BCG-Refractory Bladder Cancer; High-Risk NMIBC; Micropapillary Variant Urothelial Carcinoma (Favorable Subtype)
Keywords: Non-Muscle Invasive Bladder Cancer (NMIBC); Urothelial Carcinoma; Carcinoma in Situ (CIS); High-Grade Papillary Bladder Tumors; BCG-Unresponsive Bladder Cancer; Intravesical Chemotherapy; Gemcitabine; Docetaxel; Sequential Gemcitabine and Docetaxel; Bladder-Sparing Therapy; Radical Cystectomy Alternative; Prospective Cohort Study; Recurrence-Free Survival; Progression-Free Survival; Cystectomy-Free Survival; Cancer-Specific Survival; Quality of Life (QoL); FDA-Defined BCG Unresponsive Criteria; ECOG Performance Status; Multicenter International Trial; Bladder Preservation
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms; Carcinoma, Transitional Cell; Carcinoma in Situ | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (Experimental): High-grade non-muscle-invasive bladder cancer (HG NMIBC) with carcinoma in situ (CIS), either as pure CIS or concurrent with papillary tumors.
  Interventions: Drug: Intravesical Gemcitabine and Docetaxel
- Arm B (Experimental): High-grade non-muscle-invasive bladder cancer (HG NMIBC) with high-grade papillary tumors (stages Ta and/or T1) without carcinoma in situ (CIS).
  Interventions: Drug: Intravesical Gemcitabine and Docetaxel

INTERVENTIONS:
Drug: Intravesical Gemcitabine and Docetaxel — Sequential intravesical administration of Gemcitabine (1000mg) followed by Docetaxel (37 mg), delivered via sterile urethral catheter. Each drug is retained in the bladder for 60 minutes per instillation. The treatment consists of a 6-week induction phase (weekly instillations), followed by a 24-month maintenance phase (monthly instillations). This regimen is designed for patients with BCG-unresponsive non-muscle invasive bladder cancer (NMIBC), including carcinoma in situ (CIS) and high-grade papillary tumors (Ta/T1). The study evaluates efficacy, tolerability, and bladder preservation outcomes.

SUMMARY:
The goal of this clinical trial is to learn whether a combination of two chemotherapy drugs, Gemcitabine and Docetaxel, can treat high-grade non-muscle-invasive bladder cancer (HG-NMIBC) in adults whose cancer failed conventional BCG therapy. The drugs are given directly into the bladder (intravesically), one immediately after the other.

The study will also assess the safety of this treatment.

The main questions it aims to answer are:

Can this drug combination effectively treat HG-NMIBC that did not respond to BCG and help prevent the cancer from coming back, offering long-term protection? What side effects or medical issues do participants experience during treatment?

Researchers will evaluate this non-surgical approach as a potential alternative to bladder removal surgery (radical cystectomy), with the goal of validating it as a bladder-sparing option in this setting.

Participants will:

* Go through a screening process, including tumor removal and imaging tests
* Receive weekly bladder treatments with Gemcitabine followed by Docetaxel for 6 weeks
* If the cancer responds, continue with similar once monthly treatments (maintenance therapy) for up to 2 years
* Attend regular check-ups, including bladder exams, urine tests, biopsies, and optional quality-of-life surveys
* Possibly receive a second 6-week treatment cycle if the cancer returns early
* Be followed for up to 5 years to monitor long-term outcomes

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of intravesical sequential Gemcitabine and Docetaxel in patients with BCG-unresponsive, high-grade, non-muscle-invasive bladder cancer (HG-NMIBC). Efficacy will be measured by the complete response (CR) rate at approximately 3 months for patients with carcinoma in situ (CIS), and by the disease-free rate from high-grade disease at 3 months for patients with high-grade papillary Ta/T1 disease. CR will be confirmed through cystoscopy, urine cytology, and bladder biopsy. Disease-free rate in patients with high-grade papillary disease will be assessed by non-positive cytology and the absence of visible tumor (biopsy optional).

Two distinct patient cohorts will be recruited for this trial:

Arm A: Patients with CIS, either alone or with concurrent papillary tumors Arm B: Patients with high-grade papillary tumors (Ta and/or T1) without CIS

Secondary objectives include characterizing the safety and toxicity profile of the treatment and evaluating additional efficacy outcomes such as high-grade recurrence-free survival (HGRFS), recurrence-free survival (RFS), progression-free survival (PFS), cystectomy-free survival (CFS), cancer-specific survival (CSS), overall survival (OS), and quality of life (QoL).

The study will also assess outcomes in patients who experience early bladder cancer recurrence without progression and undergo a second 6-week induction cycle.

This is a prospective, two-arm, multicenter cohort study conducted nationally and internationally. Participants will receive intravesical Gemcitabine immediately followed by Docetaxel once weekly for 6 weeks (induction phase), followed by similar once monthly treatments for up to 24 months (maintenance phase). Patients will be followed for up to 5 years to assess long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed diagnosis of urothelial carcinoma of the bladder without synchronous or metachronous upper tract involvement or prostatic urethral involvement. Subjects with negative upper tract imaging within 6 months of the study start and visually normal prostates are potentially eligible. Those with a history of suspicious upper tract cytology or suspicious prostatic urethra visually will require additional upper tract washes and/or biopsies to rule out concurrent extravesical disease.

Eligible bladder cancer presentations include:

* Carcinoma in situ (CIS), with or without non-muscle-invasive stage Ta or T1 tumors of any grade.
* High-Grade Papillary tumors (stages Ta and/or T1) without CIS.
* All visible bladder tumors must be completely resected within 8 weeks prior to initiating intravesical Gem/Doce therapy.
* If more than 8 weeks have passed since diagnosis or resection of index bladder CIS ± non-invasive tumor (pTa or T1 tumors), an office cystoscopy must be performed within 8 weeks of Gem/Doce initiation to confirm no visible tumor regrowth.

BCG-Unresponsive Disease as defined by any of the following FDA-accepted criteria:

* Occurrence of high-grade, stage T1 cancer after at least 5/6 weekly BCG induction treatments.
* Occurrence of CIS within 12 months, or high-grade papillary disease, stage Ta/T1, within 6 months after an "adequate" course of BCG therapy.

An "adequate" course of BCG includes at least 5/6 weekly BCG induction treatments and at least 2/3 weekly BCG maintenance or 2/6 weekly BCG re-induction treatments.

* N.B: Physician may have some flexibility (+/- 1 month) in the use of 6 and 12 months to define BCG-unresponsive NMIBC.
* N.B: Once a patient has been correctly defined as having BCG-unresponsive disease, they will be considered to always be BCG-unresponsive for the purpose of this study. In other words, there is no restriction as to when the BCG-unresponsive term was assigned.

  * The occurrence of low-grade (LG) Ta disease will not be considered a HG relapse event given its prognosis is much more favorable that HG disease. However, all LG tumor must be completely resected before continuing with Gemcitabine/Docetaxel therapy.
  * Subjects must be eligible for radical cystectomy and decline this standard of care treatment or not be a surgical candidate for radical cystectomy (as appropriate) based on other comorbidities.
  * All grossly visible disease in the bladder must be fully resected with pathologic stage and grade assessed at the local study institution. Local pathologists are strongly encouraged to use the current LG and HG AJCC criteria.

NB: For institutions that still use the 3-tiered grading system, Ta Gr1 and Gr 2 will be considered LG while any Ta Gr3 or T1 Gr2 or Gr3 will be considered HG.

* Patients enrolled in other clinical trials must have received their last treatment at least 8 weeks prior to enrollment if the treatment was an intravesical agent. If the treatment included a systemic immune-modulating agent (e.g. anti-PD(L)-1 or anti CTLA4) then at least two dosing intervals must have elapsed untreated before the patient is eligible.
* Age > 18 and must be able to read, understand and sign the local informed consent.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance Status of 2 or less, including patients who are not surgical candidates due to comorbid conditions.
* Women of childbearing potential must have a negative pregnancy test at screening.
* All patients of childbearing potential must be willing to consent to using effective contraception, i.e., IUD, Birth control pills, Depo-Provera, and/or condoms while on treatment and for 3 months after their last Gemcitabine/Docetaxel treatment.
* No intravesical or upper tract topical therapy within 8 weeks of study entry.
* Must be willing and able to comply with all protocol requirements.
* Should have a Complete Blood Count (CBC) with differential before the index tumor resection or biopsy (within 30 days) and/or within 14 days before starting Gemcitabine/Docetaxel therapy.
* Must be willing and able to give informed consent and any authorizations required by the local Institutional Review Board (IRB) for participation in this study.

Exclusion Criteria:

* History or concurrent Stage T2 or greater urothelial cancer.
* History or concurrent upper tract or prostatic urethral cancer (no suspicious or positive upper tract cytology and negative upper tract imaging within 6 months of study entry; visually normal or absent prostatic urethra by cystoscopy).
* History or concurrent variant bladder cancer histology including squamous cell carcinoma, adenocarcinoma, small cell carcinoma, plasmacytoid carcinoma, nested urothelial carcinoma, sarcomatoid carcinoma, squamous, glandular, metastatic carcinoma and others. Select urothelial carcinoma with favorable micropapillary differentiation is permitted (see above).
* Active other malignancies excluding indolent or well-controlled prostate cancer, basal or squamous cell skin cancers or non-invasive cancer of the cervix are permitted so long as they are not expected to impact 3-year survival outcomes.
* History of severe hypersensitivity reaction (>= grade 3) to Gemcitabine and/or Docetaxel.
* History of severe hypersensitivity reaction (>= grade 3) to Polysorbate 80 containing drugs (Docetaxel is formulated with Polysorbate 80)
* Concurrent treatment with any intravesical or systemic chemotherapeutic agent (8-week washout required).
* Treatment with a checkpoint inhibitor within 2 treatment cycles of enrollment.
* Major surgery within 3 months of enrollment.
* Inadequate organ and bone marrow function as evidenced by:

  1. Hemoglobin ≤8.0 g/dL.
  2. Absolute neutrophil count ≤1.5 x 109/L.
  3. Platelet count ≤80 x 109/L.
  4. AST/SGOT and/or ALT/SGPT ≥3.0 x ULN.
  5. Total bilirubin >1.5 x ULN excepting known benign Gilbert's Disease.
  6. Serum creatinine >2.0 x ULN.

  i. If creatinine 1.5 - 2.0 x ULN, creatinine clearance will be calculated according to CKD-EPI formula and patients with creatinine clearance <30 mL/min should be excluded.
* History of radiation to the pelvis.
* History of difficult catheterization that in the opinion of the Investigator will prevent safe and/or reliable administration of the intravesical agents.
* History of interstitial cystitis or current inability to hold ~ 2 ounces of fluid in the bladder for the expected 60-minute retention time (assistive medication and/or techniques (gravity reflux; split dosing) are permitted).
* Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy (3- week documented clearance required).
* Known human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C infection.
* Recent Covid infection within 30 days of enrollment or currently symptomatic of Covid-related illnesses.
* Significant cardiovascular risk (e.g., coronary stenting within 8 weeks, myocardial infarction within 6 months).
* Women who are pregnant or lactating.
* Participation in any other research protocol involving administration of an investigational agent within 6 weeks of study entry (8-week washout required)
* Any other major or unstable medical condition that in the Investigator's opinion, could affect patient performance status, ability to receive the intravesical therapy and/or life expectancy during the five years of intended study participation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2033-01-01 (Estimated); Study Completion 2033-01-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Intravesical Gemcitabine/Docetaxel in BCG-Unresponsive Carcinoma In Situ NMIBC | 3 months
  To determine the efficacy of intravesical Gemcitabine/Docetaxel in patients with BCG-unresponsive carcinoma in situ (CIS) urothelial bladder carcinoma, as measured by the complete response (CR) rate (%) at approximately 3 months. CR will be determined through mandatory cystoscopy, urine cytology, and biopsy for those with CIS.
Efficacy of Intravesical Gemcitabine/Docetaxel in BCG-Unresponsive Papillary NMIBC | 3 months
  To determine the efficacy of intravesical Gemcitabine/Docetaxel in patients with BCG-unresponsive papillary urothelial bladder carcinoma, as measured by high-grade recurrence-free survival (HG RFS) rate (%) at approximately 3 months. Non-positive cytology and non-suspicious visual cystoscopic findings will determine lack of HG disease for subjects entering this study with papillary tumors (HG Ta T1).

SECONDARY OUTCOMES:
Long-Term Efficacy of Intravesical Sequential Gemcitabine/Docetaxel in BCG-Unresponsive NMIBC | Up to 60 months (5 years) from initiation of treatment, with key evaluations at 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, and 60 months
  To assess duration of complete response for CIS +/- papillary TaT1 in month
Long-Term Efficacy of Intravesical Sequential Gemcitabine/Docetaxel in BCG-Unresponsive NMIBC | Up to 60 months (5 years) from initiation of treatment, with key evaluations at 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, and 60 months
  To assess high-grade recurrence-free survival (HGRFS) for HG papillary only TaT1 in month
Long-Term Efficacy of Intravesical Sequential Gemcitabine/Docetaxel in BCG-Unresponsive NMIBC | Up to 60 months (5 years) from initiation of treatment, with key evaluations at 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, and 60 months
  To assess recurrence-free survival (RFS) in month
Long Term Efficacy of Intravesical Sequential Gemcitabine/Docetaxel in BCG-Unresponsive NMIBC | Up to 60 months (5 years) from initiation of treatment, with key evaluations at 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, and 60 months
  To assess progression-free survival (PFS) in month
Long-Term Efficacy of Intravesical Sequential Gemcitabine/Docetaxel in BCG-Unresponsive NMIBC | Up to 60 months (5 years) from initiation of treatment, with key evaluations at 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, and 60 months
  To assess cystectomy-free survival (CFS) in month
Long-Term Efficacy of Intravesical Sequential Gemcitabine/Docetaxel in BCG-Unresponsive NMIBC | Up to 60 months (5 years) from initiation of treatment, with key evaluations at 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, and 60 months
  To assess cancer-specific survival (CSS) in month
Long-Term Efficacy of Intravesical Sequential Gemcitabine/Docetaxel in BCG-Unresponsive NMIBC | Up to 60 months (5 years) from initiation of treatment, with key evaluations at 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, and 60 months
  To assess overall survival in month

OTHER OUTCOMES:
Safety of Intravesical Sequential Gemcitabine/Docetaxel in BCG-Unresponsive NMIBC: Adverse Event Analysis | Up to 60 months (5 years) from initiation of treatment, with key evaluations at 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, and 60 months
  To assess the incidence (%) of adverse events
Safety of Intravesical Sequential Gemcitabine/Docetaxel in BCG-Unresponsive NMIBC: Adverse Event Analysis | Up to 60 months (5 years) from initiation of treatment, with key evaluations at 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, and 60 months
  To assess the severity of adverse events (Common Terminology Criteria for Adverse Events (CTCAE)) (Grade I-IV)
Change in Health-Related Quality of Life Measured by FACT-Bladder (FACT-Bl) | Up to 60 months (5 years), with assessments at baseline, Week 6 of induction, and at key evaluation points: 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, and 60 months.
  The Functional Assessment of Cancer Therapy-Bladder (FACT-Bl) is a validated, patient-reported outcome measure assessing health-related quality of life in bladder cancer. It includes the FACT-G core domains: Physical Well-Being (PWB), Social/Family Well-Being (SWB), Emotional Well-Being (EWB), Functional Well-Being (FWB) plus a Bladder Cancer Subscale (BLCS). Score (range: 0-160). Higher scores indicate better quality of life.
Change in Health-Related Quality of Life Measured by FACT-General (FACT-G) | Up to 60 months (5 years), with assessments at baseline, Week 6 of induction, and at key evaluation points: 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, and 60 months.
  The Functional Assessment of Cancer Therapy-General (FACT-G) is a validated, oncology-generic patient-reported outcome covering Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, and Functional Well-Being. Total Score Range: 0-108; higher scores indicate better quality of life.
Change in Health-Related Quality of Life Using EQ-5D™ | Up to 60 months (5 years), with assessments at baseline, Week 6 of induction, and at key evaluation points: 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, and 60 months.
  EQ-5D™ is a validated instrument assessing five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. It includes a descriptive system and a visual analog scale (VAS). Index Score (U.S. value set): Range -0.573 to 1.000; higher scores indicate better health status.
  VAS: Range 0-100; higher scores indicate better perceived health
High-Grade Disease-Free Rate (HG-DFR) in Patients Re-Induced With Gemcitabine/Docetaxel After Recurrence | Up to 60 months (5 years) from initiation of treatment, with key evaluations at 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, and 60 months
  To determine the efficacy of intravesical sequential Gemcitabine/Docetaxel in patients re-induced after recurrence of BCG-unresponsive non-muscle invasive bladder cancer (NMIBC), as measured by the high-grade disease-free rate (HG-DFR, %) at prespecified time points.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A O'Donnell, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
At this time, there are no plans to share individual participant data (IPD) due to institutional data governance policies, privacy considerations, and the absence of a formal data-sharing infrastructure. Requests for data may be considered on a case-by-case basis following study completion and publication.

REFERENCES:
- [Background] Ben-David R, Tillu N, Alerasool P, Bieber C, Ranti D, Tolani S, Eisenhauer J, Chung R, Lavallee E, Waingankar N, Attalla K, Wiklund P, Mehrazin R, Anderson CB, Sfakianos JP. Induction and maintenance of sequential intravesical gemcitabine/docetaxel for intermediate and high-risk non-muscle invasive bladder cancer with different dosage protocols. World J Urol. 2024 May 11;42(1):315. doi: 10.1007/s00345-024-04992-5. PMID 38734774
- [Background] Daniels MJ, Barry E, Milbar N, Schoenberg M, Bivalacqua TJ, Sankin A, Kates M. An evaluation of monthly maintenance therapy among patients receiving intravesical combination gemcitabine/docetaxel for nonmuscle-invasive bladder cancer. Urol Oncol. 2020 Feb;38(2):40.e17-40.e24. doi: 10.1016/j.urolonc.2019.07.022. Epub 2019 Aug 28. PMID 31473090
- [Background] McElree IM, Mott SL, O'Donnell MA, Packiam VT. Alternative instillation techniques of sequential intravesical gemcitabine and docetaxel for non-muscle-invasive bladder cancer. BJU Int. 2024 Jun;133(6):671-673. doi: 10.1111/bju.16208. Epub 2023 Oct 26. No abstract available. PMID 37858923
- [Background] Alghafees M, Chakra MA, Alkhayal A, Moussa M, Alkhamees M, Alsaikhan B, Alasker A, Alsayyari A, Alsaghyir A, Alkahtani A, O'Donnell MA. Saudi urologists' treatment pattern for high-risk Bacillus Calmette-Guerin naive and Bacillus Calmette-Guerin unresponsive nonmuscle invasive bladder cancer. Urol Ann. 2025 Jan-Mar;17(1):58-63. doi: 10.4103/ua.ua_43_24. Epub 2025 Jan 18. PMID 40051987
- [Background] Abou Chakra M, Shore ND, Dillon R, O'Donnell MA. US Clinical Practice Patterns of Intravesical Chemotherapy for Bacillus Calmette-Guerin-Unresponsive and Bacillus Calmette-Guerin-Exposed Nonmuscle-Invasive Bladder Cancer. Urol Pract. 2024 Jan;11(1):97-107. doi: 10.1097/UPJ.0000000000000481. Epub 2023 Oct 30. PMID 37903746
- [Background] Abou Chakra M, Packiam VT, Duquesne I, Peyromaure M, McElree IM, O'Donnell MA. Combination intravesical chemotherapy for non-muscle invasive bladder cancer (NMIBC) as first-line or rescue therapy: where do we stand now? Expert Opin Pharmacother. 2024 Feb;25(2):203-214. doi: 10.1080/14656566.2024.2310073. Epub 2024 Jan 30. PMID 38264853
- [Background] McElree IM, Steinberg RL, Mott SL, O'Donnell MA, Packiam VT. Comparison of Sequential Intravesical Gemcitabine and Docetaxel vs Bacillus Calmette-Guerin for the Treatment of Patients With High-Risk Non-Muscle-Invasive Bladder Cancer. JAMA Netw Open. 2023 Feb 1;6(2):e230849. doi: 10.1001/jamanetworkopen.2023.0849. PMID 36853609
- [Background] Yim K, Melnick K, Mott SL, Carvalho FLF, Zafar A, Clinton TN, Mossanen M, Steele GS, Hirsch M, Rizzo N, Wu CL, Mouw KW, Wszolek M, Salari K, Feldman A, Kibel AS, O'Donnell MA, Preston MA. Sequential intravesical gemcitabine/docetaxel provides a durable remission in recurrent high-risk NMIBC following BCG therapy. Urol Oncol. 2023 Nov;41(11):458.e1-458.e7. doi: 10.1016/j.urolonc.2023.06.018. Epub 2023 Sep 9. PMID 37690933
- [Background] Chevuru PT, McElree IM, Mott SL, Steinberg RL, O'Donnell MA, Packiam VT. Long-term follow-up of sequential intravesical gemcitabine and docetaxel salvage therapy for non-muscle invasive bladder cancer. Urol Oncol. 2023 Mar;41(3):148.e1-148.e7. doi: 10.1016/j.urolonc.2022.10.030. Epub 2022 Nov 28. PMID 36456454
- [Background] Steinberg RL, Thomas LJ, Brooks N, Mott SL, Vitale A, Crump T, Rao MY, Daniels MJ, Wang J, Nagaraju S, DeWolf WC, Lamm DL, Kates M, Hyndman ME, Kamat AM, Bivalacqua TJ, Nepple KG, O'Donnell MA. Multi-Institution Evaluation of Sequential Gemcitabine and Docetaxel as Rescue Therapy for Nonmuscle Invasive Bladder Cancer. J Urol. 2020 May;203(5):902-909. doi: 10.1097/JU.0000000000000688. Epub 2019 Dec 10. PMID 31821066
- [Background] Balar AV, Kamat AM, Kulkarni GS, Uchio EM, Boormans JL, Roumiguie M, Krieger LEM, Singer EA, Bajorin DF, Grivas P, Seo HK, Nishiyama H, Konety BR, Li H, Nam K, Kapadia E, Frenkl T, de Wit R. Pembrolizumab monotherapy for the treatment of high-risk non-muscle-invasive bladder cancer unresponsive to BCG (KEYNOTE-057): an open-label, single-arm, multicentre, phase 2 study. Lancet Oncol. 2021 Jul;22(7):919-930. doi: 10.1016/S1470-2045(21)00147-9. Epub 2021 May 26. PMID 34051177
- [Background] Brahmer JR, Long GV, Hamid O, Garon EB, Herbst RS, Andre T, Armand P, Bajorin D, Bellmunt J, Burtness B, Choueiri TK, Cohen EEW, Diaz LA Jr, Shitara K, Kulkarni G, McDermott D, Shah M, Tabernero J, Vogel A, Zinzani PL, Jafari N, Bird S, Snyder E, Gause C, Bracco OL, Pietanza MC, Gruber T, Ribas A. Safety profile of pembrolizumab monotherapy based on an aggregate safety evaluation of 8937 patients. Eur J Cancer. 2024 Mar;199:113530. doi: 10.1016/j.ejca.2024.113530. Epub 2024 Jan 11. PMID 38295556
- [Background] Cookson MS, Chang SS, Lihou C, Li T, Harper SQ, Lang Z, Tutrone RF. Use of intravesical valrubicin in clinical practice for treatment of nonmuscle-invasive bladder cancer, including carcinoma in situ of the bladder. Ther Adv Urol. 2014 Oct;6(5):181-91. doi: 10.1177/1756287214541798. PMID 25276228
- [Background] Narayan VM, Boorjian SA, Alemozaffar M, Konety BR, Shore ND, Gomella LG, Kamat AM, Bivalacqua TJ, Montgomery JS, Lerner SP, Busby JE, Poch M, Crispen PL, Steinberg GD, Schuckman AK, Downs TM, Mashni J Jr, Lane BR, Guzzo TJ, Bratslavsky G, Karsh LI, Woods ME, Brown G, Canter D, Luchey A, Lotan Y, Inman BA, Williams MB, Cookson MS, Chang SS, Sankin AI, O'Donnell MA, Sawutz D, Philipson R, Parker NR, Yla-Herttuala S, Rehm D, Jakobsen JS, Juul K, Dinney CPN. Efficacy of Intravesical Nadofaragene Firadenovec for Patients With Bacillus Calmette-Guerin-Unresponsive Nonmuscle-Invasive Bladder Cancer: 5-Year Follow-Up From a Phase 3 Trial. J Urol. 2024 Jul;212(1):74-86. doi: 10.1097/JU.0000000000004020. Epub 2024 May 5. PMID 38704840
- [Background] Necchi A, Roumiguie M, Kamat AM, Shore ND, Boormans JL, Esen AA, Lebret T, Kandori S, Bajorin DF, Krieger LEM, Niglio SA, Uchio EM, Seo HK, de Wit R, Singer EA, Grivas P, Nishiyama H, Li H, Baranwal P, Van den Sigtenhorst-Fijlstra M, Kapadia E, Kulkarni GS. Pembrolizumab monotherapy for high-risk non-muscle-invasive bladder cancer without carcinoma in situ and unresponsive to BCG (KEYNOTE-057): a single-arm, multicentre, phase 2 trial. Lancet Oncol. 2024 Jun;25(6):720-730. doi: 10.1016/S1470-2045(24)00178-5. Epub 2024 May 10. PMID 38740030
- [Background] Steinberg G, Bahnson R, Brosman S, Middleton R, Wajsman Z, Wehle M. Efficacy and safety of valrubicin for the treatment of Bacillus Calmette-Guerin refractory carcinoma in situ of the bladder. The Valrubicin Study Group. J Urol. 2000 Mar;163(3):761-7. PMID 10687972
- [Background] Al Hussein Al Awamlh B, Chang SS. Novel Therapies for High-Risk Non-Muscle Invasive Bladder Cancer. Curr Oncol Rep. 2023 Feb;25(2):83-91. doi: 10.1007/s11912-022-01350-9. Epub 2022 Dec 26. PMID 36571706
- [Background] Shabsigh A, Korets R, Vora KC, Brooks CM, Cronin AM, Savage C, Raj G, Bochner BH, Dalbagni G, Herr HW, Donat SM. Defining early morbidity of radical cystectomy for patients with bladder cancer using a standardized reporting methodology. Eur Urol. 2009 Jan;55(1):164-74. doi: 10.1016/j.eururo.2008.07.031. Epub 2008 Jul 18. PMID 18675501
- [Background] Novara G, Catto JW, Wilson T, Annerstedt M, Chan K, Murphy DG, Motttrie A, Peabody JO, Skinner EC, Wiklund PN, Guru KA, Yuh B. Systematic review and cumulative analysis of perioperative outcomes and complications after robot-assisted radical cystectomy. Eur Urol. 2015 Mar;67(3):376-401. doi: 10.1016/j.eururo.2014.12.007. Epub 2015 Jan 2. PMID 25560798
- [Background] Chang SS, Boorjian SA, Chou R, Clark PE, Daneshmand S, Konety BR, Pruthi R, Quale DZ, Ritch CR, Seigne JD, Skinner EC, Smith ND, McKiernan JM. Diagnosis and Treatment of Non-Muscle Invasive Bladder Cancer: AUA/SUO Guideline. J Urol. 2016 Oct;196(4):1021-9. doi: 10.1016/j.juro.2016.06.049. Epub 2016 Jun 16. PMID 27317986
- [Background] Holzbeierlein JM, Bixler BR, Buckley DI, Chang SS, Holmes R, James AC, Kirkby E, McKiernan JM, Schuckman AK. Diagnosis and Treatment of Non-Muscle Invasive Bladder Cancer: AUA/SUO Guideline: 2024 Amendment. J Urol. 2024 Apr;211(4):533-538. doi: 10.1097/JU.0000000000003846. Epub 2024 Jan 24. PMID 38265030
- [Background] Broughton EI, Chun DS, Gooden KM, Mycock KL, Rajkovic I, Taylor-Stokes G. Treatment and disease management patterns for bacillus Calmette-Guerin unresponsive nonmuscle invasive bladder cancer in North America, Europe and Asia: A real-world data analysis. Curr Urol. 2022 Sep;16(3):147-153. doi: 10.1097/CU9.0000000000000072. Epub 2022 Aug 2. PMID 36204362
- [Background] Broughton EI, Gooden KM, Mycock KL, Rajkovic I, Taylor-Stokes G. Multi-country clinical practice patterns, including use of biomarkers, among physicians' treatment of BCG-unresponsive non-muscle invasive bladder cancer (NMIBC). BMC Urol. 2022 Feb 26;22(1):27. doi: 10.1186/s12894-022-00959-z. PMID 35219307
- [Background] Collacott H, Krucien N, Heidenreich S, Catto JWF, Ghatnekar O. Patient Preferences for Treatment of Bacillus Calmette-Guerin-unresponsive Non-muscle-invasive Bladder Cancer: A Cross-country Choice Experiment. Eur Urol Open Sci. 2023 Jan 31;49:92-99. doi: 10.1016/j.euros.2022.12.016. eCollection 2023 Mar. PMID 36874596
- [Background] Moussa M, Abou Chakra M, Shore ND, Papatsoris A, Farahat Y, O'Donnell MA. Patterns of treatment of high-risk BCG-unresponsive non-muscle invasive bladder cancer (NMIBC) patients among Arab urologists. Arch Ital Urol Androl. 2024 Mar 19;96(1):12244. doi: 10.4081/aiua.2024.12244. PMID 38502039
- [Background] Joudi FN, Smith BJ, O'Donnell MA, Konety BR. Contemporary management of superficial bladder cancer in the United States: a pattern of care analysis. Urology. 2003 Dec;62(6):1083-8. doi: 10.1016/s0090-4295(03)00765-9. PMID 14665360
- See also: Center for Biologics Evaluation and Research. (n.d.). Adstiladrin. U.S. Food and Drug Administration — https://www.fda.gov/vaccines-blood-biologics/cellular-gene-therapy-products/adstiladrin
- See also: Center for Drug Evaluation and Research. (n.d.). Drug trials snapshots: Anktiva. U.S. Food and Drug Administration. — https://www.fda.gov/drugs/drug-approvals-and-databases/drug-trials-snapshots-anktiva